CLINICAL TRIAL: NCT00406172
Title: Intravitreal Bevacizumab (Avastin) for Pseudophakic Macular Edema (PME)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: APEC 0016
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Cystoid Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab

SUMMARY:
To report safety and efficacy of intravitreal injection of bevacizumab in patients with cystoid macular edema secondary to cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pseudophakic eyes with macular edema

Exclusion Criteria:

* Other retinopathies

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Cubas-Lorenzo, MD, Principal Investigator — APEC México
Locations (1):
- APEC, México D.F., Mexico